CLINICAL TRIAL: NCT02246010
Title: Does Intake of Lactose-free Milk in Infants With Acute Gastroenteritis in a Developing Country Shorten the Duration of Diarrhea? A Randomized Clinical Trial.
Brief Title: Lactose-free Milk in Infants With Acute Diarrhea in a Developing Country
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very slow recruitment rate. Only 6 infants were recruited over 2 years.
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Mona Nabulsi, Professor of Clinical Pediatrics, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED.MN.09
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Acute Gastroenteritis
Keywords: diarrhea; developing world; lactose-free diet; Clinical trial
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactose-free milk (Experimental): Lactose- free milk formula (Similac LF®) and anti-diarrheic diet for 7 days.
  Interventions: Dietary Supplement: Lactose- free milk
- Regular infant milk (No Intervention): Regular infant milk formula and anti-diarrheic diet for 7 days.

INTERVENTIONS:
Dietary Supplement: Lactose- free milk — Lactose- free milk
  Arms: Lactose-free milk

SUMMARY:
The purpose of this study is to determine whether lactose-free milk will shorten the diarrhea duration and decrease its severity in formula-fed infants presenting to the Emergency Department (ED) or pediatric clinics with acute diarrhea.

DETAILED DESCRIPTION:
Acute gastroenteritis is a major cause of pediatric morbidity and mortality accounting for 15 % of all childhood death worldwide, and is a major public health burden, especially in developing countries. A recent Cochrane review of 33 randomized or quasi-randomized trials reported a modest reduction in the duration of diarrhea in children younger than 5 years who were on reduced or lactose-free diet. Those trials however were conducted on inpatients in high or middle-income countries. None were from developing countries where diarrheal diseases are severer and result in higher morbidities and mortalities. This study aims at investigating the effect of lactose-free milk on the duration and severity of diarrhea in infants from a developing country, who present with acute gastroenteritis to the Emergency Department (ED) or pediatric clinics. The findings from this study will help provide evidence-based dietary recommendations for infants with acute diarrhea in developing countries who are treated in the ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Infants on artificial milk formula
* Presenting to the ED or pediatric clinics of the American University of Beirut Medical Center
* Chief complaint: acute gastroenteritis (three or more loose or liquid stools in 24 hours, for at least 24 hours, and not exceeding 2 weeks from presentation, with or without fever, vomiting, mucus or blood per stools).

Exclusion Criteria:

* Exclusively or partially breast-fed infants
* Severe dehydration requiring hospitalization

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

REFERENCES:
- [Derived] Nabulsi M, Yazbeck N, Charafeddine F. Lactose-free milk for infants with acute gastroenteritis in a developing country: study protocol for a randomized controlled trial. Trials. 2015 Feb 8;16:46. doi: 10.1186/s13063-015-0565-9. PMID 25771831

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactose-free Milk | Regular Infant Milk
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Infants between 2 months and 18 months presenting with acute diarrhea.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactose-free Milk | Regular Infant Milk | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Customized [Count of Participants; unit: Participants]
  Less than 6 months | 1 | 0 | 1
  Equal or more than 6 months | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Diarrhea duration [Mean (Standard Deviation); unit: Days] — Number of days with diarrhea.
  Days | 4.2 (2.2) | 3.5 (0.7) | 4.0 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Diarrhea Duration
Description: number of days with 3 or more loose or watery stools
Time Frame: From onset of illness till the day of last diarrheic stool passed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lactose-free Milk | Regular Infant Milk
Number analyzed (Participants) | 4 | 2
Days | 8.7 (2.2) | 8.5 (2.1)

2. Secondary Outcome: Weight Loss
Description: Percent weight loss from baseline
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: percent of body weight in kilogram
Arm/Group | Lactose-free Milk | Regular Infant Milk
Number analyzed (Participants) | 4 | 2
percent of body weight in kilogram | 8.6 (0.2) | 2.5 (0.1)

3. Secondary Outcome: Illness Visits
Description: Number of participants with illness visits
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lactose-free Milk | Regular Infant Milk
Number analyzed (Participants) | 4 | 2
Participants | 3 | 1

4. Secondary Outcome: Hospitalization Rate
Description: Rate of hospitalization
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lactose-free Milk | Regular Infant Milk
Number analyzed (Participants) | 4 | 2
Participants | 0 | 0

5. Secondary Outcome: Parental Satisfaction
Description: Parental satisfaction with treatment on a Likert scale from 0 (not satisfied) to 10 (very satisfied).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lactose-free Milk | Regular Infant Milk
Number analyzed (Participants) | 4 | 2
units on a scale | 7.7 (0.6) | 9.5 (0.7)

ADVERSE EVENTS:
Time Frame: Within 7 days from enrollment.
Arm/Group | Lactose-free Milk | Regular Infant Milk
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT02246010/Prot_SAP_000.pdf